CLINICAL TRIAL: NCT02523105
Title: Evaluation of Use of Brain Activity Monitoring for Early Identification of Pharmaceutical Treatment Efficacy and Development of Depression Deterioration Events.
Brief Title: Evaluation of Use of Brain Activity Monitoring for Evaluation of Depression Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brainmarc Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0010-15; NCT02583724 (obsolete NCT alias)
Record Dates: First submitted 2015-08-10; First posted 2015-08-14 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2016-07

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Participants diagnosed with depression. (Other): EEG monitoring and evaluation
  Interventions: Device: EEG monitoring
- Healthy participants. (Other): EEG monitoring and evaluation
  Interventions: Device: EEG monitoring

INTERVENTIONS:
Device: EEG monitoring — EEG evaluation will be done using two off the shelf EEG devices for research and consumer use. The first one is a device called MindWave by NeuroSky ltd (http://neurosky.com) the second called EPOC by Emotiv ltd (https://emotiv.com/epoc.php).
  EEG evaluation will be conducted for a total duration of 20 minutes with and without auditory stimulation. The auditory stimulation will be performed using standard headphone or earphones to reduce external noises.

SUMMARY:
This study evaluates the use of brain activity monitoring for early identification of pharmaceutical treatment efficacy and development of depression deterioration events.

DETAILED DESCRIPTION:
The study will be conducted in two arms:

In arm I, participants diagnosed with depression. In arm II, healthy participants.

Arm I - Participants that need to start or switch their pharmacological antidepressant therapy will be recruited. Their clinical status will be evaluated and their EEG characteristics will be collected.

Arm II - Clinical and EEG characteristics of Healthy volunteers will collected on a similar timetable.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 -70 years (Adult, Senior)
* Able and willing to comply with all study requirements.

Additional Inclusion Criteria for Arm I

* Diagnosed with depression
* Being within 2 days of receiving pharmaceutical treatment for depression for the first

time or changing dose or changing type of current pharmaceutical treatment or addition to

drug of current pharmaceutical treatment.

Additional Inclusion Criteria for Arm II

Brief Symptom Inventory (BSI < 2.3).

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Diagnosed with Psychotic disorder.
* Diagnosed with Central Neurological disorder.
* A user of recreational or illicit drugs or has had a recent history of drug or alcohol abuse

or dependence.

* Hearing disorder and/or known ear drum impairment.
* High suicide risk as judged by the research team.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-10-09 (Actual); Study Completion 2017-01-05 (Actual)

PRIMARY OUTCOMES:
Tuning and evaluation of use of EEG analysis of brain prefrontal activity for mental status evaluation. | 12 months
  Outcome measures: optimal EEG device, sampling duration, frequency, and EEG measure dynamics correlation with depression clinical dynamics.

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Bloch, MD, Principal Investigator — Shalvata Hospital
Locations (2):
- Israel (2):
  - Haemek medical center, Afula
  - Shalvata Hospital, Hod HaSharon

REFERENCES:
- See also: A Pilot Study of Possible Easy-to-Use Electrophysiological Index for Early Detection of Antidepressive Treatment Non-Response — https://www.frontiersin.org/articles/10.3389/fpsyt.2017.00128/full